CLINICAL TRIAL: NCT04440280
Title: Targeting Reactive Oxygen Species Production as a Novel Therapeutic in Fuch's Endothelial Corneal Dystrophy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Ula Jurkunas, Associate Professor, Harvard Medical School, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P001909
Record Dates: First submitted 2020-06-11; First posted 2020-06-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Fuchs Endothelial Corneal Dystrophy
Keywords: Fuchs; Fuchs Endothelial Corneal Dystrophy; oxidative stress; N-Acetylcysteine ophthalmic drops; Descemet Membrane Endothelial Keratoplasty; DMEK
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — Acetylcysteine; Solutions

STUDY DESIGN:
Intervention Model Description: Initially, 30 eyes from up to 30 participants will be randomized 1:1 to one of two groups, a group administering N-acetyl cysteine (NAC) 10% and a group administering Visine Tears Dry Eye Relief artificial tears ophthalmic solution (the placebo).
  After interim analysis of the study with 30 eyes, if a significant difference in the primary endpoint between NAC 10% and placebo is not found, an additional 15 eyes from up to 15 participants will be enrolled to investigate 20% NAC.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind trial, where neither the study participant nor the investigators will know to which treatment group the study participant has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- NAC 10% group (Active Comparator): Subjects in this group will be treated with eye drops containing a 10% solution of N-acetyl cysteine. Topical NAC is a well-tolerated medication that has many applications in ophthalmology including dry eye disease and meibomian gland dysfunction.
  Interventions: Drug: N-acetyl cysteine (NAC) 10% solution
- NAC 20% group (Active Comparator): Subjects in this group will be treated with eye drops containing a 20% solution of N-acetyl cysteine. Topical NAC is a well-tolerated medication that has many applications in ophthalmology including dry eye disease and meibomian gland dysfunction.
  Interventions: Drug: N-acetyl cysteine (NAC) 20% solution
- Placebo group (Placebo Comparator): Subjects in this group will be treated with a placebo (Visine Tears Dry Eye Relief artificial tears ophthalmic solution.)
  Interventions: Drug: Visine Dry Eye Relief eye drops

INTERVENTIONS:
Drug: N-acetyl cysteine (NAC) 10% solution — N-acetyl cysteine is a sterile, unpreserved eye drop containing 10% (100 mg/mL) of acetylcysteine.
  Other Names: acetylcysteine
  Arms: NAC 10% group
Drug: N-acetyl cysteine (NAC) 20% solution — N-acetyl cysteine is a sterile, unpreserved eye drop containing 20% (200 mg/mL) of acetylcysteine.
  Other Names: acetylcysteine
  Arms: NAC 20% group
Drug: Visine Dry Eye Relief eye drops — Visine Tears Dry Eye Relief artificial tears ophthalmic solution
  Arms: Placebo group

SUMMARY:
This protocol will investigate whether topical application of N-acetyl cysteine (NAC) eye drops decreases oxidative stress and confers cytoprotection in patients with FECD.

DETAILED DESCRIPTION:
Fuchs Endothelial Corneal Dystrophy (FECD) is the most common corneal endothelial disorder and has been estimated to affect approximately 4% of the US population over the age of 40. Corneal transplantation is currently the primary treatment modality available to treat FECD, and there are no medical therapies that treat the disease or stall its progression. Therefore, there is an unmet need to identify pharmacotherapeutic interventions that would prevent the endothelial cell loss in early through late stages of FECD, as well as after corneal transplantation, aiding in the survival of the corneal grafts.

The investigators know that cell loss in FECD is caused by increased oxidative stress in the CEC and aqueous humor of FECD. The investigators have in vitro and in vivo data showing that the processes involved in the development of FECD can be arrested with administration of N-acetyl cysteine (NAC). Currently topical solutions of NAC are already used in ophthalmology for application in keratoconjunctivitis sicca (using 20% weight/volume solution or 10%), meibomian gland dysfunction (using 5%) and Sjögren's dry eye syndrome (also using 5%).

This is a single center, double-blind, placebo-controlled, randomized trial. Adult participants with advanced FECD and cataracts who qualify for the standard treatment (combined Descemet Membrane Endothelial Keratoplasty (DMEK) and cataract surgery) will be enrolled at Massachusetts Eye and Ear.

After meeting eligibility criteria and completing informed consent, 30 eyes from up to 30 participants with advanced FECD and cataracts with indication for combined DMEK and cataract surgery will be initially enrolled. (NOTE: Some participants may be enrolled twice if they elect to have both eyes treated within the study.) Eyes will be randomized 1:1 to NAC 10% and the placebo, Visine Tears Dry Eye Relief artificial tears ophthalmic solution. Each participant will self-administer 1 drop of study drug four times a day in the planned operative eye for 28 days prior to planned surgery.

After interim analysis of the study with 30 eyes, if a significant difference in the primary endpoint between NAC 10% and placebo is not found, an additional 15 eyes from up to 15 participants will be enrolled and assigned to 20% NAC.

Prior to and after using the study medication, participants will complete patient-reported visual disability questionnaires and have corneal measurements and images taken. Participants additionally will complete a tolerability and medication adherence questionnaire after using the study medication.

In the operating room, a standard incision will be made to collect the fluid from the anterior part of the eye and replaced with a salt solution or viscous agent routinely used during the surgery. This procedure is routinely performed during this type of surgery, however, some of the aqueous fluid will be collected and analyzed rather than being discarded. Additionally, corneal tissue which is normally removed during corneal transplantation surgery and discarded will be kept for further research on FECD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥21 years of age at time of surgical evaluation.
2. Diagnosis of advanced FECD and visually significant cataract
3. Indication for DMEK (Descemet Membrane Endothelial Keratoplasty) with concurrent cataract surgery
4. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
5. Willingness and ability to adhere to medication regimen

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
2. History of prior intraocular surgery in study eye including cataract, glaucoma and/or retina surgery
3. History of other corneal diseases, such as severe dry eye, corneal scars, pseudophakic bullous keratopathy, corneal degenerations, corneal infections
4. Use of ocular prescription medications except for lubricants, hyperosmotic agents, or ocular hypotensive agents
5. History of ocular surface infection within the past 30 days
6. Use of systemic, inhalational, or topical N-Acetylcysteine within the past 30 days
7. History of intolerance to topical N-Acetylcysteine
8. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

   -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Level of H2O2 in the aqueous humor | DMEK Surgery occurs 28 to 42 days after participant enrollment
  The primary endpoint is the level of H2O2 in the aqueous humor obtained at time of DMEK surgery.

SECONDARY OUTCOMES:
Assessment of safety of NAC eye drops in patients with FECD by documenting the number and severity of adverse events. | Ongoing safety assessment will occur starting on the first day when subjects receive the study drug, through the pre-operative visit, surgery and post-surgical follow-up visits, a period of approximately 6-7 weeks.
  Safety assessment will be ongoing for the entire 28 days that study participants take study drug (prior to surgery) and in all post surgical follow-up visits. Assessment will be based on the number and severity of adverse events, with specific scrutiny for evidence of severe ocular adverse reactions such as ocular chemosis, severe injection, presence or worsening of corneal epithelial staining and/or epithelial defects.
Assessment of tolerability of N-acetyl cysteine drops in patients with FECD by documenting participants' reports of irritation, burning, itchiness or redness in their eyes while taking the study drug | Tolerability will be assessed after participants have taken study drug for 28 days or earlier, if the participants report difficulties tolerating the drug.
  Participants will be asked to fill out a tolerability and medication adherence questionnaire where they will rate the irritation, burning, itchiness and redness they experience after using the medication on a scale of 1 to 100.
Change in patient-reported visual disability after NAC administration | Assessed when subject starts study drug and again, 21 to 28 days later.
  Change in patient-reported visual disability will be obtained using the previously validated questionnaire, V-FUCHS instrument 10 before and after the study drug is administered. Participants will be asked how often they experience specific visual difficulties selecting from the following choices: never, rarely, sometimes, most of the time or all of the time. Participants will also be asked how much difficulty they have performing certain visual tasks. Options for the answers are: No difficulty, a little difficulty, moderate difficulty, a lot of difficulty or extreme difficulty.
Change in central corneal thickness after NAC administration | Assessed when subject starts study drug and again, 21 to 28 days later.
  Change in central corneal thickness as measured by CCT; decrease by >30 µm before and after NAC drop administration period.
Change in corneal endothelial cell counts after NAC administration | Assessed when subject starts study drug and again, 21 to 28 days later.
  Change in the number of corneal endothelial cells as determined by HRT3 with Rostock Corneal Module (Heidelberg Engineering, Heidelberg, Germany) before and after NAC drop administration period. If central counts are unattainable due to end-stage of FECD, then peripheral counts will be obtained.
Changes in corneal tomography after NAC administration | Assessed when subject starts study drug and again, 21 to 28 days later.
  Corneal tomography is a three-dimensional imaging technique that characterizes the anterior/posterior corneal surfaces. Participants will have corneal tomography twice: first before they start the study drug, and then again, 28 to 42 days later when the drug treatment has concluded. Change in corneal tomography imaging will be assessed qualitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ula Jurkunas, MD, Principal Investigator — Mass Eye and Ear
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No